CLINICAL TRIAL: NCT04126330
Title: Effect of Omega-3 and Probiotic Dietary Supplements on Elevated High Sensitivity C-reactive Protein (Hs-CRP) as a Marker of Low-grade Inflammation: Targeting Inflammation and Intestinal Barrier Function in the Elderly and Obese
Brief Title: Effect of Omega-3 and Probiotic Dietary Supplements on Elevated High Sensitivity C-reactive Protein (Hs-CRP) as a Marker of Low-grade Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: University of Hohenheim (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Robert Brummer, Professor of Gastroenterology and Clinical Nutrition, Director Nutrition-Gut-Brain Interactions Research Centre, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Provita19
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Probiotics; Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: proof-of-concept, randomized double-blinded placebo-controlled parallel study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Probiotics and Omega-3/vitamin D Supplements- Elderly (Experimental)
  Interventions: Dietary Supplement: Probiotic, Omega-3, Vitamin D supplement
- Placebo- Elderly (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Probiotics and Omega-3/vitamin D Supplements- Obese (Experimental)
  Interventions: Dietary Supplement: Probiotic, Omega-3, Vitamin D supplement
- Placebo- Obese (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic, Omega-3, Vitamin D supplement — The first supplement we would like to assess is named VNP and is composed by Omega-3 Active and vitamin D. It contains a total of 1100 mg fish oils: 640 mg Omega-3 and with 300 mg eicosapentaenoic acid (EPA), 220 mg docosahexaenoic acid (DHA) plus 200 IU Vitamin D per daily dose (2 capsules).
  The second supplement we investigate is four-strain probiotics combination based on the commercially available formulation HOWARU® by DuPont; two capsules containing 10 billion CFU total (supplied by Pfizer but manufactured by Danisco, DuPont). The probiotic specific composition, contains equal amounts of each strain per capsule (1.25 x 109 CFU each): Bifidobacterium lactis Bi-07, Lactobacillus paracasei Lpc-37, Lactobacillus acidophilus NCFM, Bifidobacterium lactis Bl-04. One capsule contains 5 billion CFU (Swedish milliards).
  Arms: Probiotics and Omega-3/vitamin D Supplements- Elderly; Probiotics and Omega-3/vitamin D Supplements- Obese
Dietary Supplement: Placebo — Placebo generated for probiotic and omega-3/vitamin D supplements
  Arms: Placebo- Elderly; Placebo- Obese

SUMMARY:
Study objectives:

Immunity, Inflammation, and Brain Function To determine the effect of supplements with probiotics, Omega-3 and Vitamin D on the inflammatory marker highly sensitive CRP (primary outcome), markers of inflammation (secondary outcome), and gastrointestinal barrier function (secondary outcome) in elderly and obese cohorts that exhibit elevated inflammation at baseline.

Mobility To determine the effect of supplements with probiotics, Omega-3 and Vitamin D on joints, bones, and muscles by means of the WOMAC questionnaire, sit/stand test (muscle function) and CTX-I (cartilage degradation) as secondary endpoints in elderly and obese cohorts that exhibit elevated inflammation at baseline.

ELIGIBILITY:
Inclusion Criteria:

* 65-80 years old for elderly arms
* 25-65 years old for obese arms
* screening hs-CRP of 1.5-6 mg/L for elderly
* screening hs-CRP of 2-10 mg/L for obese
* BMI 18.5-27 for elderly
* BMI 28-40 for obese
* Signed informed consent prior to any study related procedures
* Prospect to start the study the latest 6 weeks after the screening visit although preferably as soon as they receive the screening results
* Willing to abstain from regular consumption of probiotic supplements, products containing probiotic bacteria
* Willing to abstain from regular consumption of medication known to alter gastrointestinal functions for at least 4 weeks prior to the time of the study inclusion
* Willing to fast at least 5 hours during the sugar-permeability-test and receive a standardised breakfast (e.g. Cereal bar) or other standardised meal
* Accepting to drink at least 1.5 litres of provided water in one day, during the two time points where the sugar test is performed

Exclusion Criteria:

1. Diagnosis of type 1 and/or type 2 diabetes
2. Current or within 4 weeks use of probiotic supplement prior to inclusion
3. More than 4 hours/week exercise habits
4. Immobile, defined as the inability to participate in all study related procedures
5. Dietary intake of fatty fish, fish oils containing omega-3 or pure omega- 3 supplements more than 2 times/week
6. History of complicated gastrointestinal surgery
7. Diagnosed Inflammatory Bowel Disease (IBD)
8. Current diagnosis of psychiatric disease/s or syndromes
9. Systemic use of antibiotics and/or steroid medication in the last 4 months prior to inclusion time
10. Use of any NSAID (Non-Steroidal Anti-Inflammatory Drugs) more than 3 times a week for the last 2 months and any time 3 days prior inclusion or at any time 3 days prior the barrier function test
11. Consumption of any NSAID up until 7 days prior to inclusion
12. Any condition which could interfere with the intestinal barrier function (e.g. gluten sensitivity, lactose intolerance, celiac disease, IBS, IBD) as decided by the principal investigators´ discretion
13. Drinking more than 9 standard cups of alcohol per week and/or more than 3 standard cups of alcohol per occasion.
14. Regular smoking, use of snuff, nicotine or e-cigarette use
15. Regular use, for more than three times a week for the last 2 months and any time 7 days prior to inclusion, of medications which according to the principal investigator can have an anti-inflammatory effect or affect in any way the intestinal barrier function or have an impact on the study analysis (e.g. laxatives, anti-diarrheal, anti-cholinergic).
16. Any disorder which according to the principal investigator can have an anti-inflammatory effect and/or can affect the intestinal barrier function, or that can impact an adequate analysis of the study outcomes
17. After being included in the study, starting with a medication/treatment or medical intervention that could potentially influence the study participation and/or the study analysis (e.g. the event of a fracture)
18. Radical change in diet (e.g. becoming vegetarian or if they discover that they are lactose intolerant) during the study period
19. Allergic to fish
20. Allergic to milk- or soy protein

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
hs-CRP | baseline, 4 weeks (mid-study), 8 weeks (study end)
  Decrease in overall body inflammation measured by at least 15% reduction in hs-CRP levels in blood

CONTACTS AND LOCATIONS:
Overall Officials: Robert JM Brummer, Prof MD PhD, Principal Investigator — Örebro University, Sweden
Locations (1):
- Örebo University, Örebro, Sweden